CLINICAL TRIAL: NCT02691572
Title: Comparison Between Transversus Abdominis Plane Block and Wound Infiltration for Analgesia After Cesarean Delivery
Brief Title: Transversus Abdominis Plane Block Versus Wound Infiltration for Postcesarean Analgesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Mohamed Mohamed Tawfik, Lecturer, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R/16.01.17
Record Dates: First submitted 2016-02-16; First posted 2016-02-25 (Estimated); Results first posted 2018-10-31 (Actual); Last update posted 2018-10-31 (Actual); Status verified 2016-05

CONDITIONS: Postcesarean Analgesia
MeSH Terms: interventions — Anesthesia, Spinal; Cesarean Section; Ketorolac; Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Wound Infiltration (Active Comparator): Cesarean delivery performed under spinal anesthesia (intrathecal bupivacaine 12.5 mg and intrathecal fentanyl 15 µg). At the end of surgery, 30 mL bupivacaine 0.25% will be injected subcutaneously in the surgical wound (15 mL on the upper and lower sides) by the obstetrician before skin suturing. Sham procedure will be performed after surgery. Standard analgesia (ketorolac and paracetamol) and fentanyl patient-controlled analgesia will be administered postoperatively.
  Interventions: Procedure: Spinal anesthesia; Drug: Intrathecal bupivacaine; Drug: Intrathecal fentanyl; Procedure: Cesarean delivery; Procedure: Wound infiltration; Procedure: Sham procedure; Drug: Ketorolac; Drug: Paracetamol; Procedure: Fentanyl patient-controlled analgesia
- Transversus abdominis plane block (Experimental): Cesarean delivery performed under spinal anesthesia (intrathecal bupivacaine 12.5 mg and intrathecal fentanyl 15 µg). After completion of surgery, bilateral ultrasound-guided TAP block will be performed using 20 mL bupivacaine 0.25% on each side. Standard analgesia (ketorolac and paracetamol) and fentanyl patient-controlled analgesia will be administered postoperatively.
  Interventions: Procedure: Spinal anesthesia; Drug: Intrathecal bupivacaine; Drug: Intrathecal fentanyl; Procedure: Cesarean delivery; Procedure: Transversus abdominis plane block; Drug: Ketorolac; Drug: Paracetamol; Procedure: Fentanyl patient-controlled analgesia

INTERVENTIONS:
Procedure: Spinal anesthesia — Performed at the L3-4 or L4-5 interspace using 27- or 25-gauge spinal needle.
Drug: Intrathecal bupivacaine — Bupivacaine 12.5 mg will be administered in the subarachnoid space.
Drug: Intrathecal fentanyl — Fentanyl 15 µg will be administered in the subarachnoid space.
Procedure: Cesarean delivery — Lower segment cesarean section using the Pfannenstiel incision and exteriorization of the uterus.
Procedure: Wound infiltration — 30 mL bupivacaine 0.25% will be injected subcutaneously in the surgical wound (15 mL on the upper and lower sides) by the obstetrician before skin suturing.
  Arms: Wound Infiltration
Procedure: Sham procedure — Sham procedure will be performed after surgery by moving the ultrasound probe and pressing a covered spinal needle on both sides of the patients' abdomen.
  Arms: Wound Infiltration
Procedure: Transversus abdominis plane block — Bilateral ultrasound-guided TAP block using 20 mL bupivacaine 0.25% on each side. A 7-12 MHz linear array probe and 22-gauge needle will be used. The probe will be placed transversely above the iliac crest in the anterior axillary line and the needle will be introduced in-plane with the probe from medial to lateral.
  Arms: Transversus abdominis plane block
Drug: Ketorolac — IV ketorolac 30 mg/8 h starting at the end of surgery.
Drug: Paracetamol — Oral paracetamol 1 gm/8 h starting 4 h after surgery.
Procedure: Fentanyl patient-controlled analgesia — Intravenous fentanyl: bolus dose = 20 µg, lockout interval = 7 min, 4-h dose limit = 200 µg, with no background infusion.

SUMMARY:
The study will compare the analgesic efficacy of transversus abdominis plane block and wound infiltration in parturients undergoing cesarean delivery under spinal anesthesia.

DETAILED DESCRIPTION:
This randomized, controlled, double-blind study will be conducted on ASA physical status II parturients with full-term singleton pregnancy undergoing elective cesarean delivery under spinal anesthesia. Patients will receive either ultrasound-guided transversus abdominis plane block or wound infiltration at the end of surgery. After delivery, all patients will receive standard analgesia (intravenous ketorolac and oral paracetamol) and patient-controlled analgesia with intravenous fentanyl. Total fentanyl consumption at 24 h, pain scores at 2, 4, 6, 12, and 24 h, side effects, and patient satisfaction will be compared between the 2 groups.

ELIGIBILITY:
Inclusion Criteria:

1. American Society of Anesthesiologists physical status II
2. Full-term singleton pregnancy

Exclusion Criteria:

1. Age <19 or > 40 years
2. Height <150 cm
3. Weight <60 kg
4. Body mass index ≥40 kg/m2
5. Contraindications to spinal anesthesia (patient refusal, increased intracranial tension, coagulopathy, uncorrected hypovolemia)
6. Hypersensitivity to any of the drugs used in the study
7. Significant cardiovascular, renal, or hepatic disease
8. Known fetal abnormalities
9. Emergency situations

Ages: 19 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2016-02; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed M Tawfik, MD, Principal Investigator — Mansoura University Hospital
Locations (1):
- Department of Anesthesia, Mansoura University Hospitals, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Wound Infiltration: Cesarean delivery performed under spinal anesthesia (intrathecal bupivacaine 12.5 mg and intrathecal fentanyl 15 µg). At the end of surgery, 30 mL bupivacaine 0.25% was injected subcutaneously in the surgical wound (15 mL on the upper and lower sides) by the obstetrician before skin suturing. Sham procedure was performed after surgery. Standard analgesia (ketorolac and paracetamol) and fentanyl patient-controlled analgesia were administered postoperatively
- Transversus Abdominis Plane Block: Cesarean delivery performed under spinal anesthesia (intrathecal bupivacaine 12.5 mg and intrathecal fentanyl 15 µg). After completion of surgery, bilateral ultrasound-guided TAP block was performed using 20 mL bupivacaine 0.25% on each side. Standard analgesia (ketorolac and paracetamol) and fentanyl patient-controlled analgesia were administered postoperatively
Period: Overall Study
Arm/Group | Wound Infiltration | Transversus Abdominis Plane Block
Started | 40 | 40
Completed | 39 | 39
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Wound Infiltration | Transversus Abdominis Plane Block | Total
Number analyzed (Participants) | 39 | 39 | 78
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.2 (4.4) | 26.7 (4.1) | 26.4 (4.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 39 | 78
  Male | 0 | 0 | 0
Height [Mean (Standard Deviation); unit: cm] | 163 (6) | 162 (4) | 163 (5)
Weight [Mean (Standard Deviation); unit: kg] | 86 (13) | 81.8 (9.2) | 83.9 (11.4)
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 32.3 (3.7) | 31 (3.3) | 31.7 (3.6)
Gestational age [Median (Full Range); unit: weeks] | 38 [37 to 40] | 38 [37 to 40] | 38 [37 to 40]
Nulliparous [Count of Participants; unit: Participants] | 8 | 9 | 17

OUTCOME MEASURES:

1. Primary Outcome: Cumulative Fentanyl Dose
Time Frame: 24 h
Measure: Mean (Standard Deviation); unit: mcg
Arm/Group | Wound Infiltration | Transversus Abdominis Plane Block
Number analyzed (Participants) | 39 | 39
mcg | 157.4 (63.4) | 153.3 (68.3)

2. Secondary Outcome: Cumulative Fentanyl Dose
Time Frame: 2, 4, 6, 12 h
Reporting Status: Not Posted

3. Secondary Outcome: Time to the First Postoperative Fentanyl Administration
Time Frame: 24 h
Reporting Status: Not Posted

4. Secondary Outcome: Pain Scores at Rest and Movement
Description: Assessed using 11-point verbal rating scale (0 = no pain, 10 = the worst possible pain), at rest and movement.
Time Frame: 2, 4, 6, 12, and 24 h
Reporting Status: Not Posted

5. Secondary Outcome: Number of Patients With Nausea and/or Vomiting
Description: The occurrence of nausea and/or vomiting will be observed and recorded.
Time Frame: 24 h
Reporting Status: Not Posted

6. Secondary Outcome: Level of Sedation
Description: Assessed using a 4-point scale (1 = awake and alert, 2 = minimally sedated, responds to speech, 3 = moderately sedated, rousable by tactile stimulation, 4 = deeply sedated, rousable only with painful stimulation).
Time Frame: 24 h
Reporting Status: Not Posted

7. Secondary Outcome: Number of Patients With Pruritis
Description: The occurrence of pruritis will be assessed by yes/no question and recorded.
Time Frame: 24 h
Reporting Status: Not Posted

8. Secondary Outcome: Level of Patient Satisfaction
Description: Assessed at 24 h using a 5-point scale (1 = very unsatisfied, 2 = unsatisfied, 3 = fair, 4 = satisfied, 5 = very satisfied).
Time Frame: 24 h
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Wound Infiltration | Transversus Abdominis Plane Block
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/39
Other Adverse Events (participants affected / at risk) | 0/39 | 0/39

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes